CLINICAL TRIAL: NCT04600453
Title: Prevention of Functional and Cognitive Impairment Through a Multicomponent Exercise Program in Hospitalized Elderly: Study Protocol for a Randomized Multicenter Clinical Trial
Brief Title: Prevention of Functional and Cognitive Impairment Through a Multicomponent Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Universidad Pública de Navarra (Other); Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MULTICENAG002
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Frailty; Disability Physical; Hospital Acquired Condition
MeSH Terms: conditions — Frailty; Iatrogenic Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): Multicomponent exercise group (intervention): The intervention will consist of a multicomponent exercise training programme24, which will be composed of supervised progressive resistance exercise training, balance-training and walking for 4 consecutive days. During the training period, patients will be trained in 20 min sessions twice a day (morning and evening).
  The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individual's functional capacity, using weight machines and aiming for 2-3 sets of 8-10 repetitions at an intensity of 40-60 % of 1RMcombined with balance and gait retraining exercises that progressed in difficulty and functional exercises, such as rises from a chair. The second part of the session will consist of functional exercises such as knee extension and flexion, hip abduction, balance movements, and daily walking in the hospital.
  Interventions: Other: Physical Exercise
- Usual care group (No Intervention): Usual care

INTERVENTIONS:
Other: Physical Exercise — The intervention will consist of a multicomponent exercise training programme24, which will be composed of supervised progressive resistance exercise training, balance-training and walking for 4 consecutive days. During the training period, patients will be trained in 20 min sessions twice a day. The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individual's functional capacity, using weight machines and aiming for 2-3 sets of 8-10 repetitions at an intensity of 40-60 % of 1RM combined with balance and gait retraining exercises that progressed in difficulty and functional exercises, such as rises from a chair. The second part of the session will consist of functional exercises such as knee extension and flexion, hip abduction, balance movements, and daily walking in the hospital.
  Other Names: Multicomponent exercise intervention
  Arms: Training group

SUMMARY:
The hospitalized elderly patient is conditioned by a series of circumstances unrelated to the pathological process itself that caused hospital admission and that usually worsen the results of hospitalization. In fact, the implementation of care models different from the traditional ones has shown a clear benefit in the functional results of these patients in the short and medium term. However, the components of these models that explain these better results have not been differentially evaluated. Some examples of these circumstances are the usual orders of absolute rest without any objective criteria for patients who are able to wander, the perpetuation of continuous fluid therapy, physical and chemical restraints, unnecessary permanent probes, etc. On numerous occasions, hospitalized elderly patients spend most of their time in bed, reaching even more than 83% of bedridden compared to 4% of those who stand up or are walking. The average time that a geriatric patient walks during their hospitalization ranges from 7 to 43 minutes/day. This population, by having their functional and physiological reserve reduced, are more vulnerable to the effects, for example, of bedridden, which range from functional loss or cognitive impairment, to longer stays, mortality and institutionalization, worse emotional situation, delirium, deconditioning, aspirations, pressure ulcers, and falls, decreased caloric intake, social isolation, poorer quality of life, and greater use of health-related resources. This study is a multicenter randomized clinical trial to be conducted in the acute care for elderly (ACE) units of three tertiary hospitals in Spain - Complejo Hospitalario de Navarra (CHN), Hospital Central de la Cruz Roja de Madrid (HCCRM) and Complejo Hospitalario Universitario of Albacete (CHUA). After randomization, the research team (physiotherapist, sport science specialist and geriatrician) will together perform the baseline measurement and follow-up visits of functional, pharmacological, comorbidity and cognitive assessment, as well as of mobility and strength evaluations. The intervention will consist of a multicomponent exercise training programme, which will be composed of supervised progressive resistance exercise training, balance-training and walking for 4 consecutive days. During the training period, patients will be trained in 20 min sessions twice a day (morning and evening).

ELIGIBILITY:
Inclusion Criteria:

* > 75 years
* Barthel Index ≥60 points
* Able to ambulate (with/without assistance)
* Sing the informed consent
* Able to communicate

Exclusion Criteria:

* Expected length of stay <6 days
* Terminal illness
* Very severe cognitive decline (i.e., GDS 7)
* Uncontrolled arrhythmias, acute pulmonary embolism and myocardial infarction, or extremity bone fracture in the past 3 months.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients with change in functional and cognitive status | 3 years
  The functional capacity of participants will be evaluated by the Short Physical Performance Battery (SPPB), the total score ranging from 0 (worst) to 12 points (best) which includes balance, gait and rising from a chair test. Standing balance test consists in the ability to maintain the standing position for 10s with three different foot position: parallel, semi-tandem and tandem. Walking speed measure, the time needed to progress for 4 linear meters with patient's usual speed, assigning a different score according to speed. Chair sit-to-stand assesses the ability to stand from a chair 5 consecutive times without using arms. The SPPB test has been shown to be a valid instrument for screening frailty and predicting disability, institutionalization and mortality.

SECONDARY OUTCOMES:
Rate of changes in the quality of life | 3 years
  - Changes in the quality of life measured by the Spanish version40 of the questionnaire EuroQol-5 Dimension (EQ-5D)41. It is an instrument measures 5 dimensions health status: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated according to the following levels: a) no problems; b) some problems; c) extreme problems. Besides, it contain visual analogy scale to quantify perceived health of 0 (worst health state imaginable) to 100 (best health state imaginable).
Number of patients with delirium | 3 years
  Development of delirium as assessed with the Confusion Assessment Method (CAM); feature 1, acute onset and fluctuating course; feature 2, inattention; feature 3, disorganized thinking; and feature 4, altered level of consciousness, with diagnosis of delirium requiring the presence of features 1 and 2 and either 3 or 442.
Mortality Rate | 3 years
  3-years mortality
Total use of health-related resources | 3 years
  Number of readmissions, visits to A&E, visits to outpatient clinics

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario de Navarra. Department of Geriatrics, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Garcia-Alonso Y, Galbete A, Ramirez-Velez R, Cadore EL, Izquierdo M. Short-Term Multicomponent Exercise Impact on Muscle Function and Structure in Hospitalized Older at Risk of Acute Sarcopenia. J Cachexia Sarcopenia Muscle. 2024 Dec;15(6):2586-2594. doi: 10.1002/jcsm.13602. Epub 2024 Oct 13. PMID 39400535
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Ramirez-Velez R, Zambom-Ferraresi F, Galbete A, Cadore EL, Izquierdo M. Biological sex as a tailoring variable for exercise prescription in hospitalized older adults. J Nutr Health Aging. 2024 Nov;28(11):100377. doi: 10.1016/j.jnha.2024.100377. Epub 2024 Sep 27. PMID 39341033
- [Derived] Saez de Asteasu ML, Martinez-Velilla N, Zambom-Ferraresi F, Galbete A, Ramirez-Velez R, Cadore EL, Abizanda P, Gomez-Pavon J, Izquierdo M. Dose-Response Relationship Between Exercise Duration and Enhanced Function and Cognition in Acutely Hospitalized Older Adults: A Secondary Analysis of a Randomized Clinical Trial. Innov Aging. 2024 Jun 1;8(6):igae053. doi: 10.1093/geroni/igae053. eCollection 2024. PMID 38939651